CLINICAL TRIAL: NCT00640055
Title: Using Verbal Autopsy to Determine Cause of Stillbirths and Early Neonatal Deaths Within the NICHD Global Network
Brief Title: Verbal Autopsy to Assess Early Neonatal Death and Stillbirth
Acronym: VA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: NICHD Global Network for Women's and Children's Health (Network)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Double | Purpose: Diagnostic
Other Study IDs: CP03; U01HD040636 (NIH)
Record Dates: First submitted 2008-03-18; First posted 2008-03-20 (Estimated); Last update posted 2014-07-31 (Estimated); Status verified 2014-07

CONDITIONS: Perinatal Mortality; Cause of Neonatal Death; Cause of Stilbirth
Keywords: verbal autopsy; stillbirth; neonatal death
MeSH Terms: conditions — Perinatal Death; Stillbirth

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Coordinator (non-physician)
  Interventions: Other: Coordinator
- 2 (Placebo Comparator): Physician
  Interventions: Other: Physician-assigned cause of death

INTERVENTIONS:
Other: Coordinator — Coordinator (non-physician) assigned cause of death
  Arms: 1
Other: Physician-assigned cause of death — Physician (gold standard) cause of death
  Arms: 2

SUMMARY:
The NICHD Global Network (GN) for Women's and Children's Health Research, a multi-site, international research network, provides a unique infrastructure to implement an expanded perinatal verbal autopsy study using the FIRST BREATH trial as its platform. The FIRST BREATH trial is an ongoing study of neonatal resuscitation training in rural community settings within Global Network sites in Central Africa, Asia and Latin America.

This study uses a validated VA questionnaire to determine COD of stillbirths and early neonatal deaths among participants in the FIRST BREATH study. We propose to expand the usefulness of perinatal verbal autopsy methodology in two ways. First by assessing whether the Community Coordinator (a non-physician health worker) can assign COD with a high level of concordance comparable to a Physician Panel, and second, whether the FIRST BREATH Birth Attendant can provide as reliable perinatal information as the mother during the VA interview. Our primary hypothesis is that the COD assigned by the FIRST BREATH Community Coordinator will be the same as the COD assigned by the Physician Panel in greater than 70% of early neonatal deaths (ENDs), when both use the same VA and FIRST BREATH data.

ELIGIBILITY:
Inclusion Criteria:

* Neonatal death with 7-days or stillbirth
* Lives in study cluster

Exclusion Criteria:

* Mother died
* Delivery in hospital setting

Max Age: 7 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2007-07; Primary Completion 2008-05 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Cause of death as assigned by a Community Coordinator compared to the cause of death assigned by the physician panel | 7-days

SECONDARY OUTCOMES:
The COD for stillbirth as assigned by the Community Coordinator compared to the COD for stillbirth as assigned by the Physician Panel | 7 days
The agreement between mothers' and birth attendants' responses on selected items on the VA questionnaire (considering the mothers' response as the reference standard). | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Marion Koso-Thomas, MD, Study Director — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD); Cyril Engmann, Principal Investigator — UNC at CHapel Hill
Locations (4):
- San Carlos University, Guatemala City, Guatemala
- Aga Khan University, Karachi, Pakistan
- Kinshasa School of Public Health, Kinshasa, Republic of the Congo
- University of Zambia, Lusaka, Zambia

REFERENCES:
- See also: Global Network — http://gn.rti.org